CLINICAL TRIAL: NCT01284621
Title: Relative Bioavailability of Multiple Oral Doses of BI 10773 (25 mg) and Ramipril (5 mg) Administered Together Compared to Multiple Oral Doses of BI 10773 (25 mg) Alone and Ramipril (5 mg) Alone in Healthy Male and Female Volunteers (an Open Label, Randomised, Three Way Crossover, Clinical Phase I Study)
Brief Title: Relative Bioavailability of Empagliflozin (BI 10773) and Ramipril Administered Together Compared to Empagliflozin (BI 10773) and Ramipril Alone in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1245.45; 2010-022717-25 (EudraCT Number: EudraCT)
Record Dates: First submitted 2011-01-20; First posted 2011-01-27 (Estimated); Results first posted 2014-07-22 (Estimated); Last update posted 2014-07-22 (Estimated); Status verified 2014-06

CONDITIONS: Healthy
MeSH Terms: interventions — empagliflozin; Ramipril

ARMS (3):
- BI 10773 (Experimental): 1 tablet per days for 5 days, oral administration with 240 mL water for each treatment
  Interventions: Drug: BI 10773
- Ramipril (Other): 1 tablet on day 1 and 2 tablets per day on day 2-5, oral administration with 240 mL water for each treatment
  Interventions: Drug: Ramipril
- BI 10773 + Ramipril (Other): 1 tablet BI 10773 and 1 tablet on day 1 and 2 tablets ramipril per day on day 2-5, oral administration with 240 mL water for each treatment
  Interventions: Drug: BI 10773; Drug: Ramipril

INTERVENTIONS:
Drug: BI 10773 — medium dose, oral administration
  Arms: BI 10773 + Ramipril
Drug: Ramipril — Medium dose oral administration on day 2-5
  Arms: BI 10773 + Ramipril
Drug: BI 10773 — medium dose oral administration
  Arms: BI 10773
Drug: Ramipril — Low dose oral administration on day 1
  Arms: BI 10773 + Ramipril
Drug: Ramipril — Low dose oral administration on day 1
  Arms: Ramipril
Drug: Ramipril — Medium dose oral administration on day 2-5
  Arms: Ramipril

SUMMARY:
Primary objective:To investigate if BI 10773 affects the pharmacokinetics of ramipril and if ramipril affects the pharmacokinetics of BI 10773.

ELIGIBILITY:
Inclusion criteria:

1. healthy male and female subjects

Exclusion criteria:

1. Any relevant deviation from healthy conditions.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2011-01; Primary Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- 1245.45.1 Boehringer Ingelheim Investigational Site, Biberach, Germany

REFERENCES:
- [Derived] Macha S, Sennewald R, Rose P, Schoene K, Pinnetti S, Woerle HJ, Broedl UC. Lack of clinically relevant drug-drug interaction between empagliflozin, a sodium glucose cotransporter 2 inhibitor, and verapamil, ramipril, or digoxin in healthy volunteers. Clin Ther. 2013 Mar;35(3):226-35. doi: 10.1016/j.clinthera.2013.02.015. PMID 23497760

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This was a randomised, open-label, three period, crossover study. Each treatment period was 8 days, with drug administration on days 1 to 5, and they were separated by a washout period of at least 7 days between drug administrations of 2 subsequent treatments.
Groups:
- Empa Alone / Empa + Ramipril / Ramipril Alone: Patients were administered three treatments in the following order:
  * Empagliflozin alone
  * Empagliflozin plus Ramipril
  * Ramipril
- Empa Alone / Ramipril Alone / Empa + Ramipril: Patients were administered three treatments in the following order:
  * Empagliflozin alone
  * Ramipril
  * Empagliflozin plus Ramipril
- Ramipril Alone / Empa Alone / Empa + Ramipril: Patients were administered three treatments in the following order:
  * Ramipril
  * Empagliflozin alone
  * Empagliflozin plus Ramipril
- Ramipril Alone / Empa + Ramipril / Empa Alone: Patients were administered three treatments in the following order:
  * Ramipril
  * Empagliflozin plus Ramipril
  * Empagliflozin alone
- Empa + Ramipril / Empa Alone / Ramipril Alone: Patients were administered three treatments in the following order:
  * Empagliflozin plus Ramipril
  * Empagliflozin alone
  * Ramipril
- Empa + Ramipril / Ramipril Alone / Empa Alone: Patients were administered three treatments in the following order:
  * Empagliflozin plus Ramipril
  * Ramipril
  * Empagliflozin alone
Period: First Intervention (8 Days)
Arm/Group | Empa Alone / Empa + Ramipril / Ramipril Alone | Empa Alone / Ramipril Alone / Empa + Ramipril | Ramipril Alone / Empa Alone / Empa + Ramipril | Ramipril Alone / Empa + Ramipril / Empa Alone | Empa + Ramipril / Empa Alone / Ramipril Alone | Empa + Ramipril / Ramipril Alone / Empa Alone
Started | 3 | 4 | 4 | 4 | 4 | 4
Completed | 3 | 4 | 4 | 4 | 4 | 4
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout Period 1 (7 Days)
Arm/Group | Empa Alone / Empa + Ramipril / Ramipril Alone | Empa Alone / Ramipril Alone / Empa + Ramipril | Ramipril Alone / Empa Alone / Empa + Ramipril | Ramipril Alone / Empa + Ramipril / Empa Alone | Empa + Ramipril / Empa Alone / Ramipril Alone | Empa + Ramipril / Ramipril Alone / Empa Alone
Started | 3 | 4 | 4 | 4 | 4 | 4
Completed | 3 | 4 | 4 | 4 | 3 | 4
Not Completed | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Required unexpected medical treatment | 0 | 0 | 0 | 0 | 1 | 0
Period: Second Intervention (8 Days)
Arm/Group | Empa Alone / Empa + Ramipril / Ramipril Alone | Empa Alone / Ramipril Alone / Empa + Ramipril | Ramipril Alone / Empa Alone / Empa + Ramipril | Ramipril Alone / Empa + Ramipril / Empa Alone | Empa + Ramipril / Empa Alone / Ramipril Alone | Empa + Ramipril / Ramipril Alone / Empa Alone
Started | 3 | 4 | 4 | 4 | 3 | 4
Completed | 3 | 4 | 4 | 4 | 3 | 4
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout Period 2 (7 Days)
Arm/Group | Empa Alone / Empa + Ramipril / Ramipril Alone | Empa Alone / Ramipril Alone / Empa + Ramipril | Ramipril Alone / Empa Alone / Empa + Ramipril | Ramipril Alone / Empa + Ramipril / Empa Alone | Empa + Ramipril / Empa Alone / Ramipril Alone | Empa + Ramipril / Ramipril Alone / Empa Alone
Started | 3 | 4 | 4 | 4 | 3 | 4
Completed | 3 | 4 | 4 | 4 | 3 | 4
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Third Intervention (8 Days)
Arm/Group | Empa Alone / Empa + Ramipril / Ramipril Alone | Empa Alone / Ramipril Alone / Empa + Ramipril | Ramipril Alone / Empa Alone / Empa + Ramipril | Ramipril Alone / Empa + Ramipril / Empa Alone | Empa + Ramipril / Empa Alone / Ramipril Alone | Empa + Ramipril / Ramipril Alone / Empa Alone
Started | 3 | 4 | 4 | 4 | 3 | 4
Completed | 3 | 4 | 4 | 4 | 3 | 4
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Study Overall: A randomised, open-label, three period, crossover study. The three treatments administered were
  * Empagliflozin alone
  * Ramipril
  * Empagliflozin plus Ramipril
  Each treatment period was 8 days, with drug administration on days 1 to 5, and they were separated by a washout period of at least 7 days between drug administrations of 2 subsequent treatments.
Arm/Group | Study Overall
Number analyzed (Participants) | 23
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.0 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 8

OUTCOME MEASURES:

1. Primary Outcome: Total Empa: Area Under the Curve at Steady-state Over a Uniform Dosing Interval (AUCτ,ss)
Description: Area under the concentration-time curve of the analyte in plasma at steady-state over a uniform dosing interval τ, of empagliflozin (empa).
Time Frame: 0 hours (h), 20 minutes (min), 40 min, 1h, 1.5h, 2h, 2.5h, 3h, 4h, 6h, 8h, 10h, 12h, 24h, 36h, 48h and 72h after drug administration on day 5. In addition pre-dose samples, 5 minutes predose, were collected on days 1 to 4
Population: Pharmacokinetic (PK) set: All subjects who took at least one dose of investigational treatment and provided at least one observation for at least one primary endpoint without important protocol violations relevant to the PK evaluation.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol*h/L
Groups:
- Empa Alone: Empagliflozin 25mg (Empa) was administered once daily from day 1 to day 5.
- Empa + Ramipril: Empagliflozin 25mg (Empa) was administered once daily from day 1 to day 5. A single dose of ramipril 2.5mg was administered on day 1. Ramipril 5mg was administered once daily from day 2 to day 5.
Arm/Group | Empa Alone | Empa + Ramipril
Number analyzed (Participants) | 22 | 23
nmol*h/L | 5850 (18.1) | 5680 (16.3)
Statistical Analysis 1: Comparison: Empa Alone vs Empa + Ramipril; Test type: Non-Inferiority or Equivalence — No formal testing, investigation of relative bioavailability. Ratio calculated as empa plus ramipril divided by empa alone; ANOVA; Based on ANOVA with terms for sequence, subjects within sequence, period and treatment; Geometric mean ratio = 96.55, 90% CI 2-sided [93.05 to 100.18], Standard Deviation 7.1 — Standard deviation is actually the geometric coefficient of variation (gCV)

2. Primary Outcome: Total Empa: Maximum Measured Concentration (Cmax,ss)
Description: Maximum measured concentration of the analyte in plasma at steady-state over a uniform dosing interval, τ, of empagliflozin (empa).
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol/L
Arm/Group | Empa Alone | Empa + Ramipril
Number analyzed (Participants) | 22 | 23
nmol/L | 874 (25.9) | 911 (21.1)
Statistical Analysis 1: Comparison: Empa Alone vs Empa + Ramipril; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; ANOVA; Based on ANOVA with terms for sequence, subjects within sequence, period and treatment; Geometric mean ratio = 104.47, 90% CI 2-sided [97.65 to 111.77], Standard Deviation 13.1 — Standard deviation is actually the gCV

3. Primary Outcome: Total Ramipril: Area Under the Curve at Steady-state Over a Uniform Dosing Interval (AUCτ,ss).
Description: Area under the concentration-time curve of the analyte in plasma at steady-state over a uniform dosing interval τ, of ramipril.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Groups:
- Ramipril Alone: A single dose of ramipril 2.5mg was administered on day 1. Ramipril 5mg was administered once daily from day 2 to day 5.
Arm/Group | Ramipril Alone | Empa + Ramipril
Number analyzed (Participants) | 22 | 23
ng*h/mL | 6.59 (37.0) | 7.27 (37.8)
Statistical Analysis 1: Comparison: Ramipril Alone vs Empa + Ramipril; Test type: Non-Inferiority or Equivalence — No formal testing, investigation of relative bioavailability. Ratio calculated as empa plus ramipril divided by ramipril alone; ANOVA; Based on ANOVA with terms for sequence, subjects within sequence, period and treatment; Geometric mean ratio = 108.14, 90% CI 2-sided [100.51 to 116.35], Standard Deviation 14.0 — Standard deviation is actually the gCV

4. Primary Outcome: Total Ramipril: Maximum Measured Concentration (Cmax,ss)
Description: Maximum measured concentration of the analyte in plasma at steady-state over a uniform dosing interval, τ, of ramipril.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Ramipril Alone | Empa + Ramipril
Number analyzed (Participants) | 22 | 23
ng/mL | 8.42 (45.6) | 8.97 (53.6)
Statistical Analysis 1: Comparison: Ramipril Alone vs Empa + Ramipril; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 3, analysis 1]; ANOVA; Based on ANOVA with terms for sequence, subjects within sequence, period and treatment; Geometric mean ratio = 103.61, 90% CI 2-sided [89.73 to 119.64], Standard Deviation 28.0 — Standard deviation is actually the gCV

5. Primary Outcome: Total Ramiprilat: Area Under the Curve at Steady-state Over a Uniform Dosing Interval (AUCτ,ss).
Description: Area under the concentration-time curve of the analyte in plasma at steady-state over a uniform dosing interval τ, of ramiprilat (active metabolite of ramipril).
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Ramipril Alone | Empa + Ramipril
Number analyzed (Participants) | 22 | 23
ng*h/mL | 87.2 (15.5) | 85.1 (20.1)
Statistical Analysis 1: Comparison: Ramipril Alone vs Empa + Ramipril; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 3, analysis 1]; ANOVA; Based on ANOVA with terms for sequence, subjects within sequence, period and treatment; Geometric mean ratio = 98.67, 90% CI 2-sided [96.00 to 101.42], Standard Deviation 5.2 — Standard deviation is actually the gCV

6. Primary Outcome: Total Ramiprilat: Maximum Measured Concentration (Cmax,ss)
Description: Maximum measured concentration of the analyte in plasma at steady-state over a uniform dosing interval, τ, of ramiprilat.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Ramipril Alone | Empa + Ramipril
Number analyzed (Participants) | 22 | 23
ng/mL | 11.2 (36.8) | 10.5 (46.6)
Statistical Analysis 1: Comparison: Ramipril Alone vs Empa + Ramipril; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 3, analysis 1]; ANOVA; Based on ANOVA with terms for sequence, subjects within sequence, period and treatment; Geometric mean ratio = 98.29, 90% CI 2-sided [92.67 to 104.25], Standard Deviation 11.3 — Standard deviation is actually the gCV

7. Secondary Outcome: Empa: Predose Concentration Prior to Administration of the Nth Dose (Cpre,N)
Description: Predose concentration of the analyte in plasma prior to administration of the Nth dose, of empagliflozin.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol/L
Arm/Group | Empa Alone | Empa + Ramipril
Number analyzed (Participants) | 22 | 23
nmol/L
  Cpre,2 | 40.3 (31.0) | 38.6 (32.1)
  Cpre,3 | 45.8 (33.7) | 45.1 (30.6)
  Cpre,4 | 49.2 (29.5) | 46.4 (27.2)
  Cpre,5 | 47.8 (25.5) | 48.3 (27.9)

8. Secondary Outcome: Ramiprilat: Predose Concentration Prior to Administration of the Nth Dose (Cpre,N)
Description: Predose concentration of the analyte in plasma prior to administration of the Nth dose, of ramiprilat.
  Note, predose concentrations for ramipril were all below the limit of quantification (BLQ) and therefore the predose concentration of the analyte in plasma prior to administration of the Nth dose, of ramipril was not analysed.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Ramipril Alone | Empa + Ramipril
Number analyzed (Participants) | 22 | 23
ng/mL
  Cpre,2 | 1.03 (25.5) | 1.02 (21.7)
  Cpre,3 | 1.33 (21.9) | 1.31 (17.4)
  Cpre,4 | 1.39 (20.7) | 1.37 (17.2)
  Cpre,5 | 1.45 (23.4) | 1.44 (16.6)

9. Secondary Outcome: Time From Last Dosing to the Maximum Measured Concentration (Tmax,ss)
Description: Time from last dosing to the maximum measured concentration of the analyte in plasma at steady state.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Median (Full Range); unit: hours
Arm/Group | Empa Alone | Ramipril Alone | Empa + Ramipril
Number analyzed (Participants) | 22 | 22 | 23
hours
  Total empa | 1.02 (42.6) [0.667 to 3.00] | NA (NA) [NA to NA] — Not applicable - no ramipril in this treatment arm | 1.50 (44.7) [1.00 to 4.00]
  Total ramipril | NA (NA) [NA to NA] — Not applicable - no empagliflozin in this treatment arm | 0.333 (36.4) [0.333 to 1.00] | 0.333 (39.1) [0.333 to 1.00]
  Total ramiprilat | NA (NA) [NA to NA] — Not applicable - no empagliflozin in this treatment arm | 2.00 (23.8) [1.48 to 4.02] | 2.00 (29.4) [1.50 to 4.00]

10. Secondary Outcome: Terminal Rate Constant (λz,ss)
Description: Terminal rate constant in plasma at steady-state
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: 1/h
Arm/Group | Empa Alone | Ramipril Alone | Empa + Ramipril
Number analyzed (Participants) | 22 | 22 | 23
1/h
  Total empa | 0.055 (37.9) | NA (NA) — Not applicable - no ramipril in this treatment arm | 0.050 (37.7)
  Total ramipril | NA (NA) — Not applicable - no empagliflozin in this treatment arm | 0.261 (107) | 0.298 (118)
  Total ramiprilat | NA (NA) — Not applicable - no empagliflozin in this treatment arm | 0.0095 (24.1) | 0.0091 (32.2)

11. Secondary Outcome: Terminal Half-life (T 1/2,ss)
Description: Terminal half-life of the analyte in plasma at steady-state.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Empa Alone | Ramipril Alone | Empa + Ramipril
Number analyzed (Participants) | 22 | 22 | 23
hours
  Total empa | 12.7 (37.9) | NA (NA) — Not applicable - no ramipril in this treatment arm | 13.9 (37.7)
  Total ramipril | NA (NA) — Not applicable - no empagliflozin in this treatment arm | 2.66 (107) | 2.32 (118)
  Total ramiprilat | NA (NA) — Not applicable - no empagliflozin in this treatment arm | 73.2 (24.1) | 76.2 (32.2)

12. Secondary Outcome: Mean Residence Time (MRTpo,ss)
Description: Mean residence time of the analyte in the body after oral administration at steady-state.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Empa Alone | Ramipril Alone | Empa + Ramipril
Number analyzed (Participants) | 22 | 22 | 23
hours
  Total empa | 9.95 (18.0) | NA (NA) — Not applicable - no ramipril in this treatment arm | 9.68 (16.8)
  Total ramipril | NA (NA) — Not applicable - no empagliflozin in this treatment arm | 1.29 (54.2) | 1.42 (57.8)
  Total ramiprilat | NA (NA) — Not applicable - no empagliflozin in this treatment arm | 44.7 (29.9) | 47.1 (38.7)

13. Secondary Outcome: Apparent Clearance After Extravascular Administration (CL/Fss)
Description: Apparent clearance of the analyte in plasma after extravascular administration at steady-state.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL/min
Arm/Group | Empa Alone | Ramipril Alone | Empa + Ramipril
Number analyzed (Participants) | 22 | 22 | 23
mL/min
  Total empa | 158 (18.1) | NA (NA) — Not applicable - no ramipril in this treatment arm | 163 (16.3)
  Total ramipril | NA (NA) — Not applicable - no empagliflozin in this treatment arm | 12600 (37.0) | 11500 (37.8)
  Total ramiprilat | NA (NA) — Not applicable - no empagliflozin in this treatment arm | 955 (15.5) | 979 (20.1)

14. Secondary Outcome: Apparent Volume of Distribution During the Terminal Phase (Vz/Fss)
Description: Apparent volume of distribution at steady-state during the terminal phase λz following an extravascular dose.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L
Arm/Group | Empa Alone | Ramipril Alone | Empa + Ramipril
Number analyzed (Participants) | 22 | 22 | 23
L
  Total empa | 174 (31.8) | NA (NA) — Not applicable - no ramipril in this treatment arm | 196 (40.0)
  Total ramipril | NA (NA) — Not applicable - no empagliflozin in this treatment arm | 2910 (89.1) | 2310 (97.3)
  Total ramiprilat | NA (NA) — Not applicable - no empagliflozin in this treatment arm | 6050 (32.0) | 6460 (42.5)

15. Secondary Outcome: Clinically Relevant Abnormalities for Physical Examination, Vital Signs, ECG, Blood Chemistry and Tolerability
Description: Clinically relevant abnormalities for physical examination, vital signs, ECG, blood chemistry and assessment tolerability by the investigator. New abnormal findings or worsening of baseline conditions were reported as adverse events.
Time Frame: From drug administration until end of washout period (36 days)
Population: Treated set which included all subjects who were dispensed study medication and were documented to have taken at least one dose of investigational treatment.
Measure: Number; unit: participants
Arm/Group | Empa Alone | Ramipril Alone | Empa + Ramipril
Number analyzed (Participants) | 22 | 22 | 23
participants | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Treatment duration plus following washout period (36 days)
Arm/Group | Empa Alone | Ramipril Alone | Empa + Ramipril
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/22 | 0/23
Other Adverse Events (participants affected / at risk) | 1/22 | 3/22 | 2/23
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Empa Alone (N=22) | Ramipril Alone (N=22) | Empa + Ramipril (N=23)
Nausea (Gastrointestinal disorders) | 0 | 0 | 2
Headache (Nervous system disorders) | 1 | 3 | 0/22

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes